CLINICAL TRIAL: NCT03557593
Title: Optimizing Prescribing of Antipsychotics in Long-Term Care (OPAL): A Randomized Trial to Reduce Inappropriate Antipsychotic Prescribing in Long-Term Care
Brief Title: Optimizing Prescribing of Antipsychotics in Long-Term Care
Acronym: OPAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Consortium on Neurodegeneration in Aging (Other); Canadian Frailty Network (Other)
Responsible Party: Principal Investigator, Dr. Dallas Seitz, Principal Investigator, Associate Professor, Dept. of Psychiatry, Queen's University, Queen's University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 6017760
Record Dates: First submitted 2018-04-06; First posted 2018-06-15 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Dementia
Keywords: Antipsychotic; Nursing home; Long-term care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Randomized, stepped-wedge cluster trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Educational — Multi component educational intervention in long-term care

SUMMARY:
Inappropriate antipsychotic prescribing is a key quality indicator by which clinical outcomes might be monitored and improved in LTC. A multi component intervention to reduce inappropriate antipsychotic prescribing was evaluated in ten Canadian long-term care facilities.

DETAILED DESCRIPTION:
Increasing numbers of older adults are affected by dementia, and many will eventually reside in long-term care (LTC), where antipsychotic use is relatively common. Inappropriate antipsychotic prescribing is a key quality indicator by which clinical outcomes might be monitored and improved in LTC but limited evidence exists on the most effective strategies for reducing inappropriate antipsychotic use.

The objective of the study was to evaluate a multicomponent approach to reduce inappropriate prescribing of antipsychotics in LTC.

A prospective, randomized stepped-wedge, study design was used to evaluate the effect of the intervention in 10 LTC facilities in Canada. The intervention consisted of an educational in-service, provision of evidence-based tools to assess and monitor neuropsychiatric symptoms (NPS) and monthly interprofessional team meetings.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia
* Receiving an antipsychotic medication without a diagnosis of psychosis

Exclusion Criteria:

* Diagnoses of schizophrenia, Huntington's disease
* Presence of active hallucinations and/or delusions
* Individuals at end of live or receiving palliative care

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2016-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Percentage of long-term care residents receiving any antipsychotic without a diagnosis of psychosis | 12-months
  The proportion of long-term care residents receiving any antipsychotic without a diagnosis of psychosis is a quality indicator is used by the Canadian Institute for Health Information to determine potentially inappropriate antipsychotic use. The quality indicator is calculated using information routinely collected on Resident Assessment Index-Minimum Dataset (RAI-MDS) assessments by determining the number of individuals who received antipsychotics on one of more days in the 7 days preceding index (RAI-MDS item O4a ≥ 1). Individuals with schizophrenia, Huntington's disease, hallucinations, delusions, those with a limited life expectancy and those currently receiving palliative care are excluded from the numerator and denominator of this indicator.

SECONDARY OUTCOMES:
Worsening of behavioral symptoms | 12-months
  Proportion of residents who had one or more of the following behavioural symptoms: wandering, physically or verbally abusive, or socially inappropriate behaviours) present on their target RAI-MDS assessment than on their prior assessment.
Use of physical restraints | 12-months
  Proportion of residents in daily physical restraints as of the target RAI-MDS assessment.
Depression: Proportion of residents whose mood from symptoms of depression worsened | 12-months
  Proportion of residents whose mood from symptoms of depression worsened compared to the previous RAI-MDS assessment.
Falls: Proportion of residents experiencing a fall in the 30 day | 12-months
  Proportion of residents experiencing a fall in the 30 days preceding the RAI-MDS assessment.
Pain: Proportion of residents who had pain | 12-months
  Proportion of residents who had pain on their target RAI=MDS assessment.

IPD SHARING:
Plan to Share IPD: No